CLINICAL TRIAL: NCT06666062
Title: " EVALUATION OF LOW INTENSITY LASER BIOMODULATORY EFFECT ON CRESTAL BONE CHANGES AROUND DELAYED IMPLANTS " A Randomized Controlled Clinical Trial
Brief Title: Evaluation of the Effect of Low Level Laser Therapy on Crestal Bone Changes and Secondary Stability Around Delayed Implant
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lina Amr Talaat (Other)
Responsible Party: Sponsor-Investigator, Lina Amr Talaat, BDS, periodontology and implantology, Ain shams university Clinical demonstrator oral medicine, periodontology horus university, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1211
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Laser Effect Around Dental Implant
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group (Active Comparator)
  Interventions: Other: implant placement and low level laser therapy
- Control group (Placebo Comparator)
  Interventions: Procedure: implant placement

INTERVENTIONS:
Other: implant placement and low level laser therapy — Laser biomodulation with low level laser therapy around delayed implant
  Arms: Study group
Procedure: implant placement — Delayed implant placement restoring missed tooth
  Arms: Control group

SUMMARY:
Although implant survival and success rates are prominent, there is still progress to be made in both survival and success rates, as well as in improving implant stability at implant placement in order to accomplish osseo-integration without significantly reducing peri-implant marginal bone. Low-level laser therapy (LLLT) has been postulated in studies looking into enhancing implant stability. Understanding the effect of LLLT on bone remodeling is crucial to knowing whether LLLT will enhance implant-bone interaction. LLLT prompts vascularization of the bone defect site and also stimulates osteoblasts, which can facilitate recovery of hard tissue. In addition, it has been recently reported that LLLT has positive effects in ossification and osseo-integration of dental implants.

DETAILED DESCRIPTION:
This study will be conducted to evaluate the effects of LLLT on the crestal bone changes around dental implants.

Study Setting Faculty of Dentistry, Ain Shams University. Sample size : 24 patients are eligible to the study.

•statistical analysis : Categorical data will be represented as frequency (n) and percentage (%) and will be analyzed using chi square test. Numerical data will be explored for normality by checking the data distribution, calculating the mean and median values and using Kolmogorov-Smirnov and Shapiro-Wilk tests. If the data was found to be normal, it will be presented as mean and standard deviation values and independent t-test will be used for intergroup comparison. If the assumption of normality is violated, the data will be presented as median and range values and intergroup comparison will be done using Mann-Whitney U test and Freidman's test. The significance level will be set at P ≤0.05 for all tests. Statistical analysis will be performed with IBM® SPSS® Statistics Version 25 for Windows.

Inclusion Criteria:

1. Healthy adult patients as evidenced by Burkett's oral medicine health history questionnaire (18).
2. Both genders.
3. Age from 20 -50 years old.
4. History of extraction< 6 months.
5. Site specific upper esthetic zone from right second premolar to left second premolar.

Exclusion criteria:

1. Patients taking drugs affecting bone metabolism for the past six months. eg. cyclosporine, methotrexate, synthetic retinoids
2. Smokers
3. Pregnancy and lactation
4. Patients with periodontal or periapical infections.
5. Vertical and horizontal root fracture
6. Mentally retarded Patients.

Study procedures:

1. Randomization and allocation concealment technique: Patients will be randomly allocated according to predetermined computer-generated randomization using www.Randomizer.org
2. Details of the interventions, testing and follow up:

   * Group A test:

     10 patients will be subjected to delayed implant placement with Laser Biostimulation with Low Level Laser Therapy.
   * Group B control:

     10 patients will be subjected to conventional delayed implant placement.

Study protocol and surgical steps

1. Radiographs will be taken from all patients after an intraoral examination.
2. Following the mucosal incision, the mucoperiosteal flap will be elevated.
3. Drilling will be performed at 900 rpm in both groups. All implants will be placed with the same torque (60 rpm) by the same surgeon (15).
4. All patients receive oral hygiene and post-operative care instructions. Group A: implant placement followed by laser bio- stimulation. Group B: implant placement without further intervention.

Low Level Laser Therapy Protocol:

Group A ( Test ):

In our study we applied a red diode laser (SmartM, Lasotronix, Poland) at 635 nm wavelength with biomodulating handpiece with following set parameters for the first session of LLLT output power: 100mW handpiece diameter: 2mm spot area: 0.0314cm2 average power density: 199.04mW/cm2 continuous mode, dose: 4J per point (16J/cm2) time: 10 sec per point, 4 points (irradiation on a buccal,lingual,mesial and distal side of the alveolus/implant), and total energy per session 16J Four irradiation sessions were provided with first therapy administered immediately following osteotomy and prior to implant placement and then immediately after implant placement , and then repeated on third day, seventh day, and fourteenth day after implant placement.

Parameters for the following sessions of LLLT :

output power: 100mW handpiece diameter: 8mm spot area: 0.5024cm2 average power density: 199.04mW/cm2 continuous mode, dose: 4J per point (16J/cm2) time: 10 sec per point, 4 points (irradiation on a buccal, lingual, mesial and distal side of the alveolus/implant), and total energy per session 16J

Group B (Control):

The same procedure was followed without laser application in this group.

ELIGIBILITY:
Inclusion Criteria:

* 1- Healthy adult patients as evidenced by Burkett's oral medicine health history questionnaire (18).

  2- Both genders. 3- Age from 20 -50 years old. 4- History of extraction< 6 months. 5- Site specific upper esthetic zone from right second premolar to left second premolar.

Exclusion criteria:

1. Patients taking drugs affecting bone metabolism for the past six months. eg. cyclosporine, methotrexate, synthetic retinoids
2. Smokers
3. Pregnancy and lactation
4. Patients with periodontal or periapical infections.
5. Vertical and horizontal root fracture
6. Mentally retarded Patients.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Radiographic evaluation of crestal bone changes | 3 months

SECONDARY OUTCOMES:
Evaluation of the secondary implant stability using implant stability quotient ( ISQ ) in response to LLLT. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Lina Amr Elsayed, Principal Investigator — Ain Shams University; Lina Amr Elsayed, Master candidate, Principal Investigator — Ain Shams University
Locations (1):
- Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided